CLINICAL TRIAL: NCT02783261
Title: Prospective Study of Early Contra-lateral Liver Lobar Hypertrophy After Unilobar Y-90 Selective Internal Radiation Therapy (SIRT) in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Prospective Post Y90 Liver Hypertrophy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHF/FG526P/2013
Record Dates: First submitted 2016-05-17; First posted 2016-05-26 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma; Liver Hypertrophy
Keywords: radioembolization; hypertrophy; Y90
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post Y90 hypertrophy measurement: All prospective patients who undergo unilobar SIRT for HCC at SGH or NCC are potential candidates for this study. The study aims to recruit 25 subjects and it is anticipated that 50% will be from SGH and 50% will be from NCC
  Interventions: Other: CT volumetric measurement after Y90 radioembolization

INTERVENTIONS:
Other: CT volumetric measurement after Y90 radioembolization — Liver volume will be measure at 3 time points. All patients will undergo CT volumetry at baseline, 4-6 weeks and 8-12 weeks after SIRT. The images are then measured using a commercially available 3D software (Vital's Vitrea Advanced CT Liver Oncology package) and manually corrected, reviewed and resected by a single senior radiologist to ensure consistency in following the same anatomical landmarks.

SUMMARY:
Patients undergoing Y90 radioembolization to will be followed prospectively with CT volumetry to determine post-Y90 rate of liver hypertrophy.

DETAILED DESCRIPTION:
Study protocol: Prospective study of early contra-lateral liver lobar hypertrophy after unilobar Y-90 selective internal radiation therapy (SIRT) in patients with hepatocellular carcinoma (HCC)

All patients scheduled to undergo unilobar (Right or left) SIRT with Y-90 for HCC at the Singapore General Hospital or the National Cancer Center Singapore during the study period may be enrolled. The target sample size is 25 over 2 years

Information on baseline demographics and disease staging, as well as pre- and post-treatment tumour and liver dimensions would be prospectively obtained.

The diagnosis of HCC is made based on current accepted diagnostic criteria ie. a characteristic appearance on contrast-enhanced quadriphasic CT scan and/or MRI, raised serum AFP levels and the presence of known risk factors. The RECIST criteria will be used to evaluate tumour response and disease progression at the time of the final volume determination.

Patients scheduled for unilobar SIRT will be consented for the study and enrolled into the study.

Liver volume will be measured at 3 time points.

CT volumetry will be performed at: 1) prior to treatment; 2) 4 to 6 weeks and 3) 8 to12 weeks after SIRT.

Administration of Y90 SIRT

This is based on our current institution practice. All patients would be reviewed with regards to suitability for Y90 SIRT and given appropriate counselling and advice regarding the angiographic procedures and the Y90 SIRT procedure, including potential side-effects. The patients undergo baseline blood investigations, typically liver function tests, renal function tests as well as full blood counts and coagulation profiles. All prior imaging CT and MRI were reviewed. Mapping hepatic angiography and 99mTc-MAA (micro-aggregated albumin) injection are performed according to standard technique. Prophylactic coil embolization of vessels at risk are performed either at mapping hepatic angiography or at 90Y radioembolization, at the discretion of the interventional radiologist. The catheter tip position for 99mTc-MAA injection is decided by consensus between the interventional radiologist and nuclear medicine physician during mapping hepatic angiography. 99mTc-MAA is slowly hand-injected through the indwelling catheter. Patients are subsequently immediately transferred to the gamma-camera suite for planar liver-to-lung shunt scintigraphy and SPECT/CT of the abdomen. Y90 microspheres treatment is planned by artery-specific SPECT/CT partition modelling as described in the literature.

All treatments are planned by a team of experienced nuclear medicine physicians. Y90 SIRT is performed using resin microspheres (SIR-Spheres; Sirtex Medical Ltd.) within 2 weeks of mapping hepatic angiography. Catheter tip placement is the same as that for the 99mTc-MAA injections. In accordance with our institutional protocol, all patients are observed overnight after treatment. They are discharged the following day after Bremsstrahlung planar scintigraphy of the lung and SPECT/CT of the abdomen were performed.

Measurement of liver volume

Liver volume will be measure at 3 time points. All patients will undergo CT volumetry at baseline, 4-6 weeks and 8-12 weeks after SIRT. Multiphasic dynamic contrast-enhanced hepatic CT scans are obtained with either a Dual Source CT (Siemens Medical) or Brilliance iCT (Philips Medical System). Scans will be obtained using a standard four phase liver protocol with a multidetector CT system with at least 64-channel detectors. Contrast medium is administered to the patients for acquisition of arterial-phase and portal-venous-phase and equilibrium CT images. The CT scanning parameters included collimation of 0.625-1.2mm. The reconstructed slice thickness for the scans are 0.8 - 1.5 mm and reconstruction intervals of 0.4 - 1 mm. Reconstructed CT slices have a matrix size of 512×512 pixels. The images are then measured using a commercially available 3D software (Vital's Vitrea Advanced CT Liver Oncology package) and manually corrected, reviewed and resected by a single senior radiologist to ensure consistency in following the same anatomical landmarks. The software allows saving of the work performed in order to allow reviewing and rechecking of the final measurements.

If the patients' pretreatment CT scans were performed at SGH or NCC, they need not undergo additional baseline CT scan and volumetry may be performed on these the existing imaging data. However, they will need to undergo a baseline CT scan if the pretreatment scan was performed outside the campus.

Subsequently, the patient's will need to undergo 2 follow-up CT scans at 4 to 6 weeks and 8 to 12 weeks after administration of SIRT.

Primary outcomes:

1. The change in volume of the contralateral liver volume from baseline
2. Change in volume of the ipsilateral liver from baseline
3. HCC tumor response or progression after treatment according to RECIST criteria.

Follow-up

Other than the 2 additional follow-up CT scans, patient's will undergo follow-up as per any regular non-study patient who was treated with SIRT.

ELIGIBILITY:
Inclusion Criteria:

* All patients with HCC who are to receive SIRT

  * The diagnosis of HCC is made based on current diagnostic criteria i.e. a characteristic appearance on contrast-enhanced quadriphasic CT scan and/or MRI, raised serum AFP levels and the presence of known risk factors
* Patients with tumor confined in the right/left lobe who will receive unilobar SIRT to the right/left hepatic artery
* All adult patients above 21 are eligible for the study
* Able to provide informed consent

Patients must meet all the above inclusion criteria to be enrolled into the study

Exclusion Criteria:

Any patient with the following exclusion criteria will not be eligible for the study:

* Patients who received SIRT not confined to the left or right lobe
* Patients who received other concomitant treatment
* Patients with bilobar disease at the time of treatment

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prospective patients who undergo unilobar SIRT for HCC at SGH or NCC are potential candidates for this study. The study aims to recruit 25 subjects and it is anticipated that 50% will be from SGH and 50% will be from NCC.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
liver hypertrophy | CT volumetry will be performed at: 1) within 1 month of radioembolization; 2) 4 to 6 weeks and 3) 8 to12 weeks after SIRT.
  Primary outcomes:
  The rate of change in volume of the contralateral liver volume from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian Goh, MBBS, Principal Investigator — Singhealth Foundation
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore